CLINICAL TRIAL: NCT05397223
Title: Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Modified mRNA Vaccines Using a Systems Biology Approach in Healthy Adults
Brief Title: A Study of Modified mRNA Vaccines in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-CRID-001
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2; Seasonal Influenza; Respiratory Syncytial Virus; Cytomegalovirus
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna; Influenza vaccine; mRNA-1010; mRNA-1345; Respiratory syncytial virus; RSV Seropositive; Vaccines; mRNA-1647; Cytomegalovirus; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19; Influenza, Human; Cytomegalovirus Infections | interventions — 2019-nCoV Vaccine mRNA-1273; mRNA-1010 influenza vaccine; mRNA-1345 respiratory syncytial virus vaccine; fluad vaccine; mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: mRNA-1345 (Experimental): Participants will receive single intramuscular (IM) injection of mRNA-1345 on Day 1.
  Interventions: Biological: mRNA-1345
- Part 1: mRNA-1647 2-Dose (Experimental): Participants will receive single IM injection of mRNA-1647 on Days 1 and 57.
  Interventions: Biological: mRNA-1647
- Part 1: mRNA-1647 3-Dose (Experimental): Participants will receive single IM injection of mRNA-1647 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1647
- Part 2: mRNA-1273 (Experimental): Participants will receive single IM injection of mRNA-1273 on Day 1
  Interventions: Biological: mRNA-1273
- Part 2: mRNA-1010 (Experimental): Participants will receive single IM injection of mRNA-1010 on Day 1.
  Interventions: Biological: mRNA-1010
- Part 2: FLUAD® (Active Comparator): Participants will receive single IM injection of FLUAD® on Day 1.
  Interventions: Biological: FLUAD®

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: Part 2: mRNA-1273
Biological: mRNA-1010 — Sterile liquid for injection
  Arms: Part 2: mRNA-1010
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: Part 1: mRNA-1345
Biological: FLUAD® — adjuvanted (MF59), inactivated, quadrivalent seasonal influenza vaccine
  Arms: Part 2: FLUAD®
Biological: mRNA-1647 — Sterile lyophilized product
  Arms: Part 1: mRNA-1647 2-Dose; Part 1: mRNA-1647 3-Dose

SUMMARY:
The main goal of this study is to evaluate the safety, reactogenicity, and immunogenicity of study vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 75 years of age at the time of consent (screening visit) who, in the opinion of the investigator, are in good health based on review of medical history and physical examination performed at screening. For mRNA-1647 study arms, adults 18 to <50 years of age at the time of consent (screening visit) who, in the opinion of the investigator, are in good health based on review of medical history and physical examination performed at screening.
* Body mass index (BMI) of 18 kilograms (kg)/square meter (m^2) to 35 kg/m^2 (inclusive) at the screening visit.

Exclusion Criteria:

* Participant has had close contact to someone with confirmed SARS-CoV-2, respiratory syncytial virus (RSV), or influenza infection in the past 14 days prior to the screening visit.
* Severe allergic reaction to any component of the FLUAD vaccine (active comparator), including egg protein, or after a previous dose of any influenza vaccine.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to screening (to include any systemic corticosteroids) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Participant plans to receive any licensed or authorized vaccine, including COVID-19 influenza vaccines, within 28 days before or after any study injection.
* Participant has received a NH 2021 - 2022 or 2022-2023 seasonal influenza vaccine or any other influenza vaccine, or an experimental RSV or cytomegalovirus (CMV) vaccine, within 6 months prior to study Day 1, and/or has not completed a primary vaccination series for COVID-19.
* Participant has received an authorized or approved COVID-19 vaccine within 4 months prior to Day 1, and/or has not completed a primary vaccination series for COVID-19.
* Participant had a laboratory-confirmed infection with influenza or RSV within 6 months prior to Day 1, or SARS-CoV-2 within 4 months of Day 1. SARS-CoV-2 infection confirmed with self-administered, authorized or approved rapid antigen test is acceptable.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the screening visit or plans to donate blood products during the study.
* Participated in an interventional clinical study within 28 days prior to the screening visit based on the medical history interview or plans to do so while participating in this study until 12 months after their last study vaccination.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 176 (7 days follow-up post-vaccination)
Number of Participants With Unsolicited Adverse Events (AEs) | Up to Day 197 (28 days follow-up post-vaccination)
Number of Participants With Serious AEs (SAEs), AEs of Special Interest (AESIs), and AEs Leading to Study Withdrawal or Discontinuation of Study Vaccination | Day 1 through end of study (EOS) (up to Day 1249)
Number of Participants with Medically Attended Adverse Events (MAAEs) | Day 1 through Day 361

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum Neutralizing Antibody Response for mRNA-1010 (and Licensed Influenza Vaccine Comparator), mRNA-1273, and mRNA-1345 | Days 1 (Baseline), 29, 85, and 197
Geometric Mean Fold-Rise (GMFR) of Serum Neutralizing Antibody Response for mRNA-1010 (and Licensed Influenza Vaccine Comparator), mRNA-1273, and mRNA-1345 | Days 1 (Baseline), 29, 85, and 197
Percentage of Participants With Seroresponse for mRNA-1010 (and Licensed Influenza Vaccine Comparator), mRNA-1273, mRNA-1345, and mRNA-1647 | Days 1 (Baseline), 29, 85, and 197

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - CenExel, Hollywood, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Meridian Clinical Research, Sioux City, Iowa
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Meridian Clinical Research, Lincoln, Nebraska
  - Benchmark Research, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - DM Clinical Research- Texas Center for Drug Development, Houston, Texas

REFERENCES:
- [Derived] Henry C, Makrinos D, Liu R, Cavallaro M, Fenderson B, Sun Y, Chang X, Astley E, Girard B, Yu WH, Oostendorp J, DiPiazza A, Paris R. An mRNA influenza vaccine induces immunity comparable to an adjuvanted vaccine in a randomized trial. NPJ Vaccines. 2026 Jan 14. doi: 10.1038/s41541-026-01370-7. Online ahead of print. PMID 41535296
- [Derived] Kaplonek P, Vargas R, Lee JS, Bertera H, Astley E, Girard B, Oostendorp J, Henry C, Paris R, Yu WH, Alter G. mRNA-1010 influenza vaccine elicits distinct and enhanced humoral immunity compared to adjuvanted inactivated vaccines. NPJ Vaccines. 2025 Dec 15. doi: 10.1038/s41541-025-01340-5. Online ahead of print. PMID 41398408
- [Derived] Fierro C, Sanchez-Crespo N, Makrinos D, Zhang W, Sun Y, Rohilla P, Girard B, Adeniji A, DiPiazza A, Paris R. Shared clinical and immunologic features of mRNA vaccines: preliminary results from a comparative clinical study. Front Immunol. 2025 Apr 10;16:1501275. doi: 10.3389/fimmu.2025.1501275. eCollection 2025. PMID 40276503